CLINICAL TRIAL: NCT01102790
Title: Generation of HIT-antibodies Without Prior Heparin Exposure Following Orthopedic Surgery (Subgroup Study) (Change of Coagulation Parameters Under Exposition With New Anticoagulants [Title of the Main Study])
Brief Title: Generation of Heparin-induced Thrombocytopenia (HIT)-Antibodies Without Prior Heparin Exposure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Edelgard Lindhoff-Last, Professor, J.W.Goethe University Hospital, Department of Internal Medicine, Division of Vascular Medicine
Other Study IDs: 243/09
Record Dates: First submitted 2010-04-07; First posted 2010-04-13 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Heparin-Induced Thrombocytopenia; Thrombosis
Keywords: HIT
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum citrated blood edta blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the HIT-antibody generation without prior heparin-exposure in patients undergoing orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major orthopedic surgery

Exclusion Criteria:

* Heparin exposure
* Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a primary care clinic undergoing orthopedic surgery without heparin exposure
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
incidence of HIT-antibodies | between day 5 and day 14 after surgery

SECONDARY OUTCOMES:
thromboembolic events | up to 21 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schindewolf, MD, Principal Investigator — J.W. Goethe University-Hospital Frankfurt/M.; Edelgard Lindhoff-Last, Prof., Principal Investigator — J.W. Goethe-University Hospital Frankfurt/M.
Locations (1):
- J.W.Goethe University Hospital Frankfurt/M., Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Schindewolf M, Lindhoff-Last E. Fondaparinux-related thrombocytopenia in a patient with former HIT. Response to Rota et al. (Thromb Haemost 2008; 99: 779-781). Thromb Haemost. 2008 Jul;100(1):168-9; author reply 169-70. doi: 10.1160/TH08-04-0222. No abstract available. PMID 18612559
- [Background] Warkentin TE, Makris M, Jay RM, Kelton JG. A spontaneous prothrombotic disorder resembling heparin-induced thrombocytopenia. Am J Med. 2008 Jul;121(7):632-6. doi: 10.1016/j.amjmed.2008.03.012. PMID 18589060
- [Background] Jay RM, Warkentin TE. Fatal heparin-induced thrombocytopenia (HIT) during warfarin thromboprophylaxis following orthopedic surgery: another example of 'spontaneous' HIT? J Thromb Haemost. 2008 Sep;6(9):1598-600. doi: 10.1111/j.1538-7836.2008.03040.x. Epub 2008 May 29. No abstract available. PMID 18513213